CLINICAL TRIAL: NCT03018275
Title: Beginning Assessment of Cutaneous Treatment Efficacy of Roseomonas in Atopic Dermatitis Phase I/II
Brief Title: Beginning Assessment of Cutaneous Treatment Efficacy of Roseomonas in Atopic Dermatitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 170033; 17-I-0033
Record Dates: First submitted 2017-01-11; First posted 2017-01-12 (Estimated); Last update posted 2019-11-27 (Actual); Status verified 2019-10

CONDITIONS: Atopic Dermatitis
Keywords: Lyophilized Biotherapeutic, Microbiome, Probiotic; Commensal Gram-negative Bacteria; Staphylococcus Aureus; Transepidermal Water Loss; Allergic Diseases
MeSH Terms: conditions — Dermatitis, Atopic; Staphylococcal Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): Vials of lyophilized R mucosa (10"3, 10"4, or 10"5 CFU)
  Interventions: Biological: Roseomonas mucosa

INTERVENTIONS:
Biological: Roseomonas mucosa — R mucosa grown in Hank's balanced salt solution. Bacteria is washed, quantitated spectrophotometrically, suspended in 10%-15% sucrose, and lyophilized.

SUMMARY:
Background:

Atopic dermatitis (AD) is a skin disease also called eczema. It is common in children and sometimes gets better on its own. However, chronic AD may cause asthma, food allergies, eye infections, and sleep problems. The cause of AD might be related to bacteria that live on the skin. Researchers want to see if introducing bacteria, R mucosa, from healthy skin onto the skin of someone with AD helps treat the disease.

Objective:

To test the safety and activity of R mucosa for treating AD.

Eligibility:

Part 1: People ages 18 and older with AD

Part 2: Children ages 3-17 with AD

Design:

Participants will be screened with:

Medical history

Physical exam

Examination of their AD

Blood and urine tests

At the baseline visit, participants will have blood tests and photos taken of their skin. They will get a supply of R mucosa and a memory aid to track their doses and record how they are feeling. Part 2 participants guardians will complete questionnaires about their child s AD.

Part 1 participants will spray R mucosa on their arm twice per week for 6 weeks.

Part 2 guardians will spray it on their child s arm twice per week for 16 weeks.

Participants will have follow-up visits to repeat some baseline tests and review their memory aid:

Part 1: Six weeks after the baseline visit

Part 2: Four times over 16 weeks; then 2 or 3 times for 1 year

Participants will be called or emailed to discuss how they are feeling:

Part 1: About 30 days after their last visit

Part 2: About every 10 days between visits

DETAILED DESCRIPTION:
The underlying pathology of atopic dermatitis (AD) consists of defective skin barrier function, susceptibility to Staphylococcus aureus skin infection, and immune imbalance. There is currently no cure for AD. Preclinical data in a mouse model of AD suggest that commensal Gram-negative bacteria (CGN), such as Roseomonas mucosa, from a healthy source can relieve symptoms of AD and have antimicrobial effects. In this study, we will first evaluate the safety of R mucosa-based biotherapy in adults with AD (age 18+ years; part 1), and then evaluate the safety and activity of R mucosa-based biotherapy in children (ages 3-17 years) with AD (parts 2A and 2B). In part 1, participants will receive twice-weekly doses of CGN biotherapy for 6 weeks, with dose escalations at 2 and 4 weeks. In part 2, participants will receive twice-weekly doses of CGN biotherapy for 4 months, with possible dose escalations at 4 and 8 weeks (part 2A only). Starting at 12 weeks for both parts 2A and 2B, dosing frequency may be increased to every other day. Participants in part 1 will be contacted 30 10 days after end of treatment for assessment of safety. Participants in parts 2A and 2B will also be followed for up to 1 year after the end of treatment for evaluation of long-term activity and safety. This will be the first study to test cutaneous live biotherapeutic products for AD. We hypothesize that altering the strains of CGN on the skin of people with AD will improve the patient s clinical outcome. We do not expect serious toxicities because R mucosa is rarely pathogenic; reported cases of bacteremia have typically been associated with percutaneous catheters in immunocompromised patients, who are excluded from this study.

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion Criteria for Young Adults and Adults with AD (Part 1)

1. Age 16+ years
2. SCORAD of at least 10
3. Have a clinical diagnosis of AD with active involvement of the antecubital fossa
4. Willing to allow storage of blood for future research
5. No history of other skin disease
6. Initiated or attempted standard of care therapy at least 6 months prior to enrollment
7. Must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) when engaging in sexual activities that can result in pregnancy. The effects of CGN live biotherapy on the developing human fetus are unknown. Adequate contraception must be used consistently, beginning before the first dose and lasting for the duration of study participation. Participants of childbearing potential must have a negative pregnancy test result before they receive CGN live biotherapy. During the course of the study, if a participant becomes pregnant or suspects they are pregnant, then they should inform the study staff and their primary care physician immediately.

Inclusion Criteria for Children with AD (Part 2)

1. Age 3-16 years
2. SCORAD of at least 10
3. Have a clinical diagnosis of AD with active involvement of the antecubital fossa
4. Willing to allow storage of blood and bacterial swabs for future research
5. Initiated or attempted standard of care therapy at least 6 months prior to enrollment
6. Participants who have begun menstruating must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) when engaging in sexual activities that can result in pregnancy.

EXCLUSION CRITERIA:

1. Presence of an indwelling venous or arterial catheter
2. Individuals living with anyone with a diagnosed immunodeficiency, cardiac valvular disease, and/of indwelling catheter
3. Precence of allergies to aimkacin, ciprofloxacin, gentamicin, levofloxacin, and tobramycin (which would preclude treatment of any unexpected infection)
4. History of cardiac valvular disease
5. Any history of grade 2 or higher neutropenia or leukopenia
6. Clinical suspicion of immunodeficiency, liver disorder, kidney disorder, and/or HIV
7. Pregnant or breastfeeding
8. Any history of anti-TNF treatment
9. Inability to demonstrate proper bacteria administration procedure despite coaching and training
10. Use of fluoroquinolone or aminoglycoside antibiotics within 2 weeks of enrollment
11. Any condition that, in the opinion of the investigator, contraindicates participation in this Study

Co-enrollment guidelines: Co-enrollment in other trials is restricted, other than enrollment on observational studies or those evaluating the use of a licensed medication. Study staff should be notified of co-enrollment as it may require the approval of the investigator.

Ages: 3 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2019-10-11 (Actual); Study Completion 2019-10-11 (Actual)

PRIMARY OUTCOMES:
A 50% reduction in antecubital-specific SCORing Atopic Dermatitis (SCORAD) with no adverse events related to product use. Frequency of solicited adverse events, unsolicited adverse events, serious adverse events, and death. | 4 weeks, 8 weeks, 12 weeks, 16 weeks, 8 months, 12 months, and 16 months

SECONDARY OUTCOMES:
A 30% improvement in the quality of life as measured by the validated Children's Dermatology Life Quality Index (CDLQI) | 4 weeks, 8 weeks, 12 weeks, 16 weeks, 8 months, 12 months, and 16 months
A 30% improvement in the quality of life as measured by the validated Family Dermatology Life Quality Index (FDLQI) | 4 weeks, 8 weeks, 12 weeks, 16 weeks, 8 months, 12 months, and 16 months

CONTACTS AND LOCATIONS:
Overall Officials: Ian A Myles, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Boguniewicz M, Leung DY. Recent insights into atopic dermatitis and implications for management of infectious complications. J Allergy Clin Immunol. 2010 Jan;125(1):4-13; quiz 14-5. doi: 10.1016/j.jaci.2009.11.027. PMID 20109729
- [Background] Myles IA, Williams KW, Reckhow JD, Jammeh ML, Pincus NB, Sastalla I, Saleem D, Stone KD, Datta SK. Transplantation of human skin microbiota in models of atopic dermatitis. JCI Insight. 2016 Jul 7;1(10):e86955. doi: 10.1172/jci.insight.86955. PMID 27478874
- [Background] Bantz SK, Zhu Z, Zheng T. The Atopic March: Progression from Atopic Dermatitis to Allergic Rhinitis and Asthma. J Clin Cell Immunol. 2014 Apr;5(2):202. doi: 10.4172/2155-9899.1000202. PMID 25419479